CLINICAL TRIAL: NCT01561079
Title: Fetal and Infant Effects of Maternal Buprenorphine Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00051600
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Buprenorphine; Methadone; Fetal neurobehavior; Infant neurobehavior
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maternal buprenorphine treatment (Experimental): Buprenorphine maintenance during pregnancy
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Daily sublingual buprenorphine treatment of pregnant, opioid dependent women from up to 34 weeks gestation through one month of infant age.
  Other Names: Subutex

SUMMARY:
This research will track the longitudinal neurobehavioral development of the buprenorphine-exposed fetus across gestation through 1 month of age in an effort to determine the safety of this medication for use during gestation, the relationship between maternal physiologic changes due to buprenorphine administration and newborn functioning, and to determine potential fetal neurobehavioral markers that may predict Neonatal Abstinence Syndrome expression and infant neurobehavioral outcome. Comparisons to results from a similar project in methadone-exposed pregnancies will be made. This proposal seeks to advance the way the investigators inform the treatment of the opioid dependent woman during pregnancy and her infant after birth.

DETAILED DESCRIPTION:
There is an increase in the prevalence of illicit opiate use among women of childbearing age in many countries today. Methadone is the treatment of choice for opioid dependency during pregnancy in the US because it markedly diminishes withdrawal symptoms and craving and blocks opioid effects, however, in utero exposure results in significant depression of fetal neurobehaviors such as fetal heart rate and heart rate variability and fetal motor activity, and significant neonatal abstinence syndrome (NAS) in the majority of exposed infants. Since its approval in 2002, the prescription of buprenorphine for opioid dependence has increased dramatically but, as with methadone, this mediation is not approved for use during pregnancy. Currently, women treated with buprenorphine prior to pregnancy are transitioned to methadone treatment due to a lack of information regarding the effects of buprenorphine on the developing fetus and infant. Pilot work by this research team suggests that buprenorphine- as compared to methadone-exposed fetuses display more optimal neurobehavioral functioning in the second and third trimesters of pregnancy. Although these results are encouraging, there is a critical need to explore fully the effects of this medication on the fetus and infant to adequately advise care providers and patients regarding its use. This is particularly true given the imminent publication of a pivotal study comparing buprenorphine to methadone treatment during pregnancy which has suggested the optimality of buprenorphine for the treatment of opioid dependence during pregnancy, and is likely to result in increasing numbers of women being treated with off-label buprenorphine during pregnancy. This proposal seeks to explore the effect of buprenorphine on maternal physiology and fetal neurobehavioral functioning longitudinally as a measure of the development of the fetal nervous system. Additionally, the neurobehavioral profile and NAS of the buprenorphine-exposed infant up to one month will be delineated in an effort to provide information necessary to provide optimal pharmacologic and non-pharmacologic treatment of NAS. Furthermore, this group has previously explored similar parameters in methadone-exposed fetuses and infants, and results of this study can be compared to those historical data. These parameters will advance our understanding of the way the investigators view and implement the future pharmacologic treatment of the opiate dependent woman during pregnancy and her infant after birth, and inform clinicians, health insurance companies and regulatory agencies in the provision of optimal care to the opioid dependent pregnant woman and her offspring before and after birth.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM) IV-R criteria
* 18-40 years of age with uncomplicated singleton pregnancies
* Accurate gestational age dating verified by ultrasound
* Gestation of less than 34 weeks
* Stabilization on buprenorphine for one week prior to study procedures

Exclusion Criteria:

* Complications of pregnancy, including gestational diabetes, polyhydramnios, hypertension, placenta previa or significant risk of preterm delivery (i.e. incompetent cervix)
* Evidence of fetal malformation detected by prenatal ultrasound
* Significant general maternal health problems that can affect fetal functioning, including Type I or gestational diabetes, alterations in thyroid functioning, HIV infection or hypertension.
* Significant maternal psychopathology that would preclude informed consent (i.e. schizophrenia)
* Alcohol dependency per DSM IV R criteria (see ascertainment methods below)
* Women stable on methadone maintenance (defined as more than 3 days of methadone dosing)
* Women entering drug treatment reporting using "street" methadone (for more than 3 days)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Center for Addiction and Pregnancy, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jansson LM, Dipietro JA, Velez M, Elko A, Williams E, Milio L, O'Grady K, Jones HE. Fetal neurobehavioral effects of exposure to methadone or buprenorphine. Neurotoxicol Teratol. 2011 Mar-Apr;33(2):240-3. doi: 10.1016/j.ntt.2010.09.003. Epub 2010 Sep 22. PMID 20868741
- [Derived] Velez ML, McConnell K, Spencer N, Montoya L, Tuten M, Jansson LM. Prenatal buprenorphine exposure and neonatal neurobehavioral functioning. Early Hum Dev. 2018 Feb;117:7-14. doi: 10.1016/j.earlhumdev.2017.11.009. Epub 2017 Dec 7. PMID 29223912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a comprehensive care treatment facility for pregnant and postpartum women with substance use disorders between Feb 2012 and March 2016
Pre-assignment Details: Participants must have an opioid use disorder, a singleton, generally uncomplicated pregnancy, be between 18 and 40 years of age, have accurate gestational age dating of less than 34 weeks, willing to receive obstetric care at the center and deliver their infant at the hospital affiliated with the treatment facility.
Groups:
- Maternal Buprenorphine Treatment: Daily sublingual buprenorphine treatment of pregnant, opioid dependent women Subjects undergo maternal-fetal monitoring at any combination of the following gestational time periods: 24, 28,32, 36 weeks of gestation
Period: Overall Study
Arm/Group | Maternal Buprenorphine Treatment
Started | 127
Completed | 49
Not Completed | 78
Not completed — Physician Decision | 17
Not completed — Withdrawal by Subject | 59
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Fetal: Daily sublingual buprenorphine treatment of pregnant, opioid dependent women Subjects completing any maternal-fetal monitoring at any combination of the following gestational ages: 24, 28, 32 36 weeks
Arm/Group | Fetal
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Education [Mean (Standard Deviation); unit: years] | 11.5 (1.9)
Age at first substance use [Mean (Standard Deviation); unit: years] | 19.8 (4.8)
Age at regular substance use [Mean (Standard Deviation); unit: years] | 21.0 (4.6)
Duration of regular substance use upon treatment entry [Mean (Standard Deviation); unit: years] | 6.5 (4.4)
Gestational age upon treatment entry [Mean (Standard Deviation); unit: weeks] | 21.3 (7.0)
Length of time in treatment prior to delivery [Mean (Standard Deviation); unit: days] | 121.1 (56.7)
Buprenorphine dose at 24 weeks if gestation [Mean (Standard Deviation); unit: mg] | 12.0 (7.1)
Buprenorphine dose at 28 weeks if gestation [Mean (Standard Deviation); unit: mg] | 12.3 (6.0)
Buprenorphine dose at 32 weeks if gestation [Mean (Standard Deviation); unit: mg] | 12.7 (6.3)
Buprenorphine dose at 36 weeks if gestation [Mean (Standard Deviation); unit: mg] | 12.8 (6.5)
Urine toxicology screenings during treatment [Mean (Standard Deviation); unit: number of screenings] | 16.4 (8.0)
Positive research urine toxicology screening at delivery [Mean (Standard Deviation); unit: percent positive urine tox. screenings] | 19.7 (25.6)

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate
Description: Fetal heart rate in beats per minute at time of trough and peak maternal buprenorphine levels
Time Frame: 24, 28, 32 and 36 weeks of gestation
Population: Participants active in the protocol at 24, 28, 32 and 36 weeks, respectively
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- FHR 24 Weeks Trough: Fetal heart rate in beats per minute at 24 weeks of gestation at trough
- FHR 28 Weeks Trough: Fetal heart rate in beats per minute at 28 weeks of gestation at time of trough maternal buprenorphine level
- FHR 32 Weeks Trough: Fetal heart rate in beats per minute at 32 weeks of gestation at time of trough maternal buprenorphine level
- FHR 36 Weeks Trough: Fetal heart rate in beats per minute at 36 weeks of gestation at time of trough maternal buprenorphine level
- FHR 24 Weeks Peak: Fetal heart rate in beats per minute at 24 weeks of gestation at time of peak maternal buprenorphine level
- FHR 28 Weeks Peak: Fetal heart rate in beats per minute at 28 weeks of gestation at time of peak maternal buprenorphine level
- FHR 32 Peak: Fetal heart rate in beats per minute at 32 weeks of gestation at time of peak maternal buprenorphine level
- FHR 36 Peak: Fetal heart rate in beats per minute at 36 weeks of gestation at time of peak maternal buprenorphine level
Arm/Group | FHR 24 Weeks Trough | FHR 28 Weeks Trough | FHR 32 Weeks Trough | FHR 36 Weeks Trough | FHR 24 Weeks Peak | FHR 28 Weeks Peak | FHR 32 Peak | FHR 36 Peak
Number analyzed (Participants) | 20 | 30 | 42 | 40 | 20 | 30 | 42 | 40
beats per minute | 145.7 (5.8) | 143.3 (5.4) | 138.6 (6.0) | 136.3 (7.1) | 143.9 (6.4) | 141.0 (4.8) | 135.4 (6.3) | 131.3 (6.1)
Statistical Analysis 1: Comparison: FHR 24 Weeks Trough vs FHR 28 Weeks Trough vs FHR 32 Weeks Trough vs FHR 36 Weeks Trough vs FHR 24 Weeks Peak vs FHR 28 Weeks Peak vs FHR 32 Peak vs FHR 36 Peak; Test type: Superiority or Other; p = 0.001, Hierarchical Linear Modeling — The p values were not adjusted for multiplicity The a priori threshold = .05; The p-value was calculated

2. Primary Outcome: Fetal Heart Rate Variability
Description: Fetal heart rate variability at 24, 28, 32 and 36 weeks of gestation at times of trough and peak maternal buprenorphine levels
Time Frame: 24, 28, 32 and 36 weeks of gestation
Population: Per protocol
Measure: Mean (Standard Deviation); unit: msec
Groups:
- FHRV 24 Trough: Fetal heart rate variability at 24 weeks of gestation at time of trough maternal buprenorphine level
- FHRV 28 Trough: Fetal heart rate variability at 28 weeks of gestation at time of trough maternal buprenorphine level
- FHRV 32 Trough: Fetal heart rate variability at 32 weeks of gestation at time of trough maternal buprenorphine level
- FHRV 36 Trough: Fetal heart rate variability at 36 weeks of gestation at time of trough maternal buprenorphine level
- FHRV 24 Peak: Fetal heart rate variability at 24 weeks gestation at the time of peak maternal buprenorphine levels
- FHRV 28 Peak: Fetal heart rate variability at 28 weeks gestation at the time of peak maternal buprenorphine levels
- FHRV 32 Peak: Fetal heart rate variability at 32 weeks gestation at the time of peak maternal buprenorphine levels
- FHRV 36 Peak: Fetal heart rate variability at 36 weeks gestation at the time of peak maternal buprenorphine levels
Arm/Group | FHRV 24 Trough | FHRV 28 Trough | FHRV 32 Trough | FHRV 36 Trough | FHRV 24 Peak | FHRV 28 Peak | FHRV 32 Peak | FHRV 36 Peak
Number analyzed (Participants) | 20 | 30 | 42 | 40 | 20 | 30 | 42 | 40
msec | 5.4 (1.3) | 6.7 (1.9) | 7.5 (3.0) | 7.9 (2.1) | 4.9 (1.5) | 7.3 (1.8) | 7.0 (2.7) | 6.3 (2.1)
Statistical Analysis 1: Comparison: FHRV 24 Trough vs FHRV 28 Trough vs FHRV 32 Trough vs FHRV 36 Trough vs FHRV 24 Peak vs FHRV 28 Peak vs FHRV 32 Peak; Test type: Superiority or Other; p < .002, Hierarchical Linear Modeling

3. Primary Outcome: Accelerations of Fetal Heart Rate
Description: Number of accelerations of fetal heart rate exhibited during the 60 minute recordings
Time Frame: 24, 28, 32 36 weeks of gestation
Measure: Mean (95% Confidence Interval); unit: accelerations
Groups:
- Accelerations 24 Trough: Accelerations in fetal heart rate at 24 weeks of gestation at time of trough maternal buprenorphine level
- Accelerations 28 Trough: Accelerations in fetal heart rate at 28 weeks of gestation at time of trough maternal buprenorphine level
- Accelerations 32 Trough: Accelerations in fetal heart rate at 32 weeks of gestation at time of trough maternal buprenorphine level
- Accelerations 36 Trough: Accelerations in fetal heart rate at 36 weeks of gestation at time of trough maternal buprenorphine level
- Accelerations 24 Peak: Accelerations in fetal heart rate at 24 weeks of gestation at time of peak maternal buprenorphine level
- Accelerations 28 Peak: Accelerations in fetal heart rate at 28 weeks of gestation at time of peak maternal buprenorphine level
- Accelerations 32 Peak: Accelerations in fetal heart rate at 32 weeks of gestation at time of peak maternal buprenorphine level
- Accelerations36 Peak: Accelerations in fetal heart rate at 36 weeks of gestation at time of peak maternal buprenorphine level
Arm/Group | Accelerations 24 Trough | Accelerations 28 Trough | Accelerations 32 Trough | Accelerations 36 Trough | Accelerations 24 Peak | Accelerations 28 Peak | Accelerations 32 Peak | Accelerations36 Peak
Number analyzed (Participants) | 20 | 30 | 42 | 40 | 20 | 30 | 42 | 40
accelerations | 0.52 [0 to 3] | 1.59 [0 to 8] | 3.57 [0 to 15] | 5.28 [0 to 17] | 0.43 [0 to 3] | 2.12 [0 to 7] | 2.29 [0 to 9] | 2.25 [0 to 9]
Statistical Analysis 1: Comparison: Accelerations 24 Trough vs Accelerations 28 Trough vs Accelerations 32 Trough vs Accelerations 36 Trough vs Accelerations 24 Peak vs Accelerations 28 Peak vs Accelerations 32 Peak vs Accelerations36 Peak; Test type: Superiority or Other; p = 0.0001, Hierarchical Linear Modeling

4. Primary Outcome: Fetal Movement
Description: Fetal movement (number x duration of fetal movements) during the 60 minute recordings at times of trough and peak maternal buprenorphine levels
Time Frame: 24, 28, 32, 36 weeks of gestation
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Fetal Movement 24 Trough; Fetal Movement 28 Trough; Fetal Movement 32 Trough; Fetal Movement 36 Trough: Fetal movement during the 60 minute recordings at 24 weeks of gestation at time of trough maternal buprenorphine level
- Fetal Movement 24 Peak; Fetal Movement 28 Peak; Fetal Movement 32 Peak; Fetal Movement 36 Peak: Fetal movement during the 60 minute recordings at 24 weeks of gestation at time of peak maternal buprenorphine level
Arm/Group | Fetal Movement 24 Trough | Fetal Movement 28 Trough | Fetal Movement 32 Trough | Fetal Movement 36 Trough | Fetal Movement 24 Peak | Fetal Movement 28 Peak | Fetal Movement 32 Peak | Fetal Movement 36 Peak
Number analyzed (Participants) | 20 | 30 | 42 | 40 | 20 | 30 | 42 | 40
seconds | 1496.2 (752.0) | 1390.0 (795.4) | 1458.7 (674.6) | 1446.7 (979.5) | 1613.0 (575.6) | 1385.7 (674.5) | 1381.2 (830.7) | 1038.2 (756.2)
Statistical Analysis 1: Comparison: Fetal Movement 24 Trough vs Fetal Movement 28 Trough vs Fetal Movement 32 Trough vs Fetal Movement 36 Trough vs Fetal Movement 24 Peak vs Fetal Movement 28 Peak vs Fetal Movement 32 Peak vs Fetal Movement 36 Peak; Test type: Superiority or Other; p = .008, Hierarchical Linear Modeling; The reported p-value was calculated

5. Primary Outcome: Fetal Movement - Fetal Heart Rate Coupling
Description: The integration between fetal movements and heart rate (FM-FHR coupling) was quantified as the proportion of time individual movements were associated with a change in FHR, using previously developed criteria. FM-FHR coupling reflects coactivation of the sympathetic and parasympathetic components of the autonomic nervous system.
Time Frame: 24, 28, 32, 36 weeks of gestation
Measure: Mean (Standard Deviation); unit: percentage of time FM assoc w FHR change
Groups:
- FM-FHR 24 Trough; FM-FHR 28 Trough; FM-FHR 32 Trough; FM-FHR 36 Trough: Fetal movement-fetal heart rate coupling during the 60 minute recordings at 24 weeks of gestation at time of trough maternal buprenorphine level
- FM-FHR 24 Peak; FM-FHR 28 Peak; FM-FHR 32 Peak; FM-FHR 36 Peak: Fetal movement-fetal heart rate coupling during the 60 minute recordings at 24 weeks of gestation at time of peak maternal buprenorphine level
Arm/Group | FM-FHR 24 Trough | FM-FHR 28 Trough | FM-FHR 32 Trough | FM-FHR 36 Trough | FM-FHR 24 Peak | FM-FHR 28 Peak | FM-FHR 32 Peak | FM-FHR 36 Peak
Number analyzed (Participants) | 20 | 30 | 42 | 40 | 20 | 30 | 42 | 40
percentage of time FM assoc w FHR change | 0.13 (0.06) | 0.21 (.07) | 0.23 (0.10) | 0.25 (0.11) | 0.09 (0.06) | 0.20 (0.09) | 0.21 (0.10) | 0.20 (0.10)
Statistical Analysis 1: Comparison: FM-FHR 24 Trough vs FM-FHR 28 Trough vs FM-FHR 36 Trough vs FM-FHR 24 Peak vs FM-FHR 28 Peak vs FM-FHR 32 Peak vs FM-FHR 36 Peak; Test type: Superiority or Other; p = .002, Hierarchical Linear Modeling

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Groups:
- Maternal Buprenorphine Treatment: Buprenorphine maintenance during pregnancy
  Buprenorphine: Daily sublingual buprenorphine treatment of pregnant, opioid dependent women from up to 34 weeks gestation through one month of infant age.
  Two severe adverse events were reported in the same infant patient. One infant had congenital heart disease and polydactyly
Arm/Group | Maternal Buprenorphine Treatment
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 1/49
Other Adverse Events (participants affected / at risk) | 15/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Buprenorphine Treatment (N=49)
Severe adverse event (Congenital, familial and genetic disorders) | 1 (1) — One infant born to a buprenorphine maintained mother in the protocol had polydactyly The infant had a family history of polydactyly
congenital heart disease (Cardiac disorders) | 1 (1) — One infant born to a buprenorphine maintained mother was born with a congenital heart disease. The infant had a family history of congenital heart disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maternal Buprenorphine Treatment (N=49)
Cholestasis of pregnancy (Hepatobiliary disorders) | 3 (3) — Three participants developed cholestasis of pregnancy. All three had concurrent Hepatitis C infection and were therefore at increased risk for this condition.
Bacterial vaginosis (Infections and infestations) | 1 (1) — One subject developed bacterial vaginosis
choroid plexus cysts (Nervous system disorders) | 1 (1) — One fetal subject had choroid plexus cysts on fetal sonogram
cardiomegaly (Cardiac disorders) | 2 (2) — 2 fetal subjects had mild cardiomegaly on fetal sonogram
pneumonia (Infections and infestations) | 1 (1) — One infant was born with congenital pneumonia
fetal growth restriction (General disorders) | 1 (1) — One fetus was diagnosed with fetal growth restriction (but was average for gestational age at delivery)
chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 2 (2) — Two maternal subjects had chorioamnionitis at delivery
Fetal stress at delivery (Pregnancy, puerperium and perinatal conditions) | 2 (2) — Two fetuses exhibited fetal stress at the time of delivery
psychiatric concern (General disorders) | 1 (1) — One maternal subject developed a psychiatric concern warranting hospitalization
fetal arrythmia (Cardiac disorders) | 1 (1) — One fetus had a cardiac arrhythmia
maternal dehydration (General disorders) | 1 (1) — One maternal subject developed decreased fetal HRV and fetal tachycardia, was dx with dehydration
nonreactive fetal tracing, fetal hear rate deceleration (Pregnancy, puerperium and perinatal conditions) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No